CLINICAL TRIAL: NCT05319158
Title: The Effect of the Movement Imitation Therapy for Preterm Babies (MIT-PB) on Motor Behavior Quality. Quasi-experimental Design.
Brief Title: The Effect of the Movement Imitation Therapy in Preterm (MIT-PB) in Motor Behavior's Quality.
Acronym: MIT-PB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Hospital Parc Taulí (Sabadell, Barcelona) (Unknown)
Responsible Party: Principal Investigator, Susana Trallero Rodríguez, PhD candidate, MsC, Physiotherapist Susana Trallero Rodríguez, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2021.002
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Premature Birth; Risk; Early Intervention
Keywords: neonatal therapy; general movements; high risk neurodevelopment; physiotherapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The infants will be pre-stratified according to General Movement Optimality Score (GMOs). The Control group will receive standard care and the Intervention groups will begin the therapy at 34-36w. The intervention will be explained and guided by the principal researcher and experienced Pediatric Physical therapist. Parents will conduct the intervention until the 50-52 weeks PMA. General Movement Assessment (GMA) will be performed at term, 44w and 54w PMA.
  Motor assessment will be carried out at 6 months Corrected Age (CA) and a global assessment at 12 months CA.
  Those assessments will be performed by independent and blind professionals at their corresponding Hospitals.
Who Masked: Outcomes Assessor
Masking Description: The assessments for the main outcome will be performed by a blinded expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The group intervention will receive MIT-PB.
  Interventions: Other: MIT-PB, movement imitation therapy for preterm.
- control group (No Intervention): The control group will receive standard care

INTERVENTIONS:
Other: MIT-PB, movement imitation therapy for preterm. — The instant an infant showed CS or PR movements, the therapists (or a therapist and a parent) intervened by gently guiding the infants' limbs so as to maneuver and smoothen their movements, thereby imitating normal GM sequences as closely as possible, adding variability to the movement
  Arms: Intervention group

SUMMARY:
This study aims to assess the effect of a parent-administered intervention program based on MIT-PB in preterm with abnormal general movements during the preterm period. We will describe the short and long-term differences between infants exposed to MIT-PB and infants who follow current standard care.

DETAILED DESCRIPTION:
The quasi-experimental design has been planned to assess the effect of a physiotherapy program carried out in neonatal intensive care and at home during the first months of life. Preterm babies born before 32 weeks gestational age (GA) and/or with less than 1500g showing an abnormal General Movement Assessment (GMA) at 34-36 weeks will be included.

Standardized tests will be performed at baseline, at term, 44 weeks post-menstrual age (PMA), 54 weeks PMA, 6 months, and 12 months.

A qualitative study has been designed to assess the physiotherapy performance and parents' experience.

Three different Hospitals with similar care protocols and sizes will recruit the sample (n=36). The Intervention groups (n=18) will be located at Hospital Josep Trueta of Girona and Hospital Sant Joan de Déu and the control group (n=18) will be located at Hospital Parc Taulí of Sabadell (Barcelona).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born before 32w GA and less than 1500g weight.
* Infants who show Abnormal General Movements (CS-PR pattern) at 34-36w postmenstrual age (PMA).
* Families able to understand/speak Catalan, Spanish or English.
* Families willing to participate who have the informed consent

Exclusion Criteria:

* Infants with congenital abnormalities and/or genetic disorders
* Infants with invasive ventilation or Continuous Positive Airway Pressure (CPAP) at 36 weeks PMA.
* Infants with Normal General Movements at 34-36 w PMA.
* Families not willing to participate.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The quality of General Movement by General Movements Optimality Score (GMOS-R) and Motor Optimality Score (MOS). | Each participant will be assessed from birth to the 54 weeks PMA.
  We will videotape General Movements at 34, 38-40, 44 and 54 weeks PMA. The baseline measure( 34w) will be performed by the main researcher and an independent and experienced certified rater. This rater will be blind regarding infant group.
  The assessments at 38-40, 44 and 54 weeks will be performed by the independent, blind and certified rater in order to guarantee the study validity.
  The GMOS-R global assessment can be Normal (N), Poor Repertoire (PR), Cramped Syncronized (CS) or Chaotic (CH). On the detailed score ,the maximum value is 38. The MOS global assessment can be classified as Fidgety (F), Abnormal Fidgety (AF) or Absent Fidgety (F-). On the detailed score the maximum value is 28. Higher scores in both scales are correlated with better global outcome.

SECONDARY OUTCOMES:
Motor development by Hammersmith Infant Neurological Scale (HINE). | 6 months CA
  Infants will assessed at 6 months CA by an independent neuro-pediatrician using the HINE.
  It is a standardized neurological exam for infants adjusted age 2 to 24 months. The HINE evaluates nerve function, movements, reflexes and reactions, posture, and tone and can help clinicians identify movement disorders including cerebral palsy (CP)The maximum global score is 78. Higher scores indicate better neurological performance.
Global development by Bayley III | 12 months CA
  An independent neuropsychologists will assess Global Development by Bayley III at 12 months CA.
  Bayley-III provides information about whether a child's developmental trajectory in the cognitive domain is proceeding as expected, relative to same-age peers. It also includes a motor score, and fine and gross motor subtest scores. The assessment indicates mild, moderate or severe delay.

OTHER OUTCOMES:
Describe families experiences with the MIT-PB | 6 months CA
  • Families will fill up a questionnaire at the end of the intervention to give their opinion about their experience with the therapy.
Study family's participation and treatment adherence | 6 months CA
  Parents will get a software application in order to register the number of treatments achieved during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Trallero, MsC, Principal Investigator — International University of Catalonia
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona, Barcelona
  - Hospital Parc Taulí de Sabadell, Sabadell, BARCELONA
  - Hospital Universitari Josep Trueta de Girona, Girona, Girona

IPD SHARING:
Plan to Share IPD: No